CLINICAL TRIAL: NCT05288140
Title: Efficacy of the Use of Diaries in Intensive Care Units
Acronym: QUADERN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Pilar Muñoz Rey, principal investigator, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PI-18-138
Record Dates: First submitted 2022-02-01; First posted 2022-03-21 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Diary (Blank Journal); Intensive Care Unit; Patient; Family; PICS; Stress; Anxiety; Depression; Quality of Life
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: A control group and an experimental group
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual ICU practice (No Intervention): The patient's evolution is reported verbally to the family.
- ICU diary (Experimental): Made a diary
  Interventions: Other: use of diary

INTERVENTIONS:
Other: use of diary — a diary is made for the experimental group where the events and events during the period of sedation and intubation are explained
  Arms: ICU diary

SUMMARY:
Randomized clinical trial that aims to evaluate the impact of the use of a diary in patients and relatives of patients admitted to an ICU in relation to usual practice in terms of health-related quality of life, the post-traumatic stress and anxiety/depression at 2, 6 and 12 months after ICU discharge.

DETAILED DESCRIPTION:
Randomized, parallel, open, non-blinded, multicenter clinical trial, with an experimental group (diary) and a control group (usual practice), to compare the effect produced on quality of life by post-traumatic stress and anxiety/depression of patients and relatives, whether or not they have access to a diary during the stay in the unit. Three validated scales will be used at three different times. 120 cases per group, carrying out a preliminary pilot test. Data analysis according to IBM SPSS v.24 to describe and compare both groups.

ELIGIBILITY:
Inclusion Criteria:

* admitted intensive care unit
* sedated and mechanically ventilated for 24hours
* signed consent
* not language barrier
* willingness to attend follow-up visits

Exclusion Criteria:

* verbal manifestation of psychiatric, mental or cognitive antecedents
* who do not coluntarily agree to participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 2 months
  questionnaries, range of 0-21 for either anxiety and depression subscores. Higher scores corresponding to worse outcomes. 0-7 normal; 8-10 borderline abnormal; 11-21 sever symptoms of anxiety or depressin.
Hospital Anxiety and Depression Scale (HADS) | 6 months
  questionnaries, range of 0-21 for either anxiety and depression subscores. Higher scores corresponding to worse outcomes. 0-7 normal; 8-10 borderline abnormal; 11-21 sever symptoms of anxiety or depressin.
Hospital Anxiety and Depression Scale (HADS) | 12 months
  questionnaries, range of 0-21 for either anxiety and depression subscores. Higher scores corresponding to worse outcomes. 0-7 normal; 8-10 borderline abnormal; 11-21 sever symptoms of anxiety or depressin.
SF-36 Health Survey | 2 months
  questionnaries to measure quality of life. 36 items. from 0 to 100, with 100 being the best health
SF-36 Health Survey | 6 months
  questionnaries to measure quality of life. 36 items. from 0 to 100, with 100 being the best health
SF-36 Health Survey | 12 months
  questionnaries to measure quality of life. 36 items. from 0 to 100, with 100 being the best health
Revised Impact of Event Scales (IES-R) | 2 months
  questionnaries; measuring areas of hyperarousal, avoidance, and intrusion as subscales. Total score ranges from 0-88, higher score associated with worse PTSD symptoms. 1-22 mild PTSD,;22 signal clinically significant PTSD symptoms.
Revised Impact of Event Scales (IES-R) | 6 months
  questionnaries; measuring areas of hyperarousal, avoidance, and intrusion as subscales. Total score ranges from 0-88, higher score associated with worse PTSD symptoms. 1-22 mild PTSD,;22 signal clinically significant PTSD symptoms.
Revised Impact of Event Scales (IES-R) | 12 months
  questionnaries; measuring areas of hyperarousal, avoidance, and intrusion as subscales. Total score ranges from 0-88, higher score associated with worse PTSD symptoms. 1-22 mild PTSD,;22 signal clinically significant PTSD symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munoz-Rey P, Romero-Garcia M, Angles-Sabate I, Ausio-Dot A, Alonso-Fernandez S, Alcala-Jimenez I, Huertas-Zurriaga A, Tur-Rubio C, Delgado-Hito P. Efficacy of the intensive care unit diary: a mixed-method study protocol. BMC Nurs. 2026 Jan 19. doi: 10.1186/s12912-026-04300-z. Online ahead of print. PMID 41555387